CLINICAL TRIAL: NCT04600843
Title: Effects of Patient Education Manual on Pain, Range of Motion and Function in Patient With Chronic Low Back Pain Neck Pain
Brief Title: Effects of Patient Education Manual in Patient With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1003 Mubashra
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Back Disorder
Keywords: Back Pain Exercise Therapy; Patient Education Manual
MeSH Terms: interventions — Physical Therapy Modalities; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy with Patient education (Experimental): Treated with proper physical therapy treatment protocol according to patient presenting condition and patient education manual
  Interventions: Other: Physical therapy with Patient education
- Physical Therapy without patient Education (Experimental): Treated with proper physical therapy treatment protocol according to patient presenting condition
  Interventions: Other: Physical Therapy without patient Education

INTERVENTIONS:
Other: Physical therapy with Patient education — patient manual was translated and validated in Urdu which was provided to patients so that they can follow it at home
  Other Names: patient education manual
  Arms: Physical therapy with Patient education
Other: Physical Therapy without patient Education — Group B was only treated with proper physical therapy treatment protocol according to patient presenting condition
  Arms: Physical Therapy without patient Education

SUMMARY:
It was a randomized clinical trial conducted to determine the effects of patient education manual on pain, range of motion and function in patient with chronic low back pain at Salamat hospital Satellite Town Gujranwala in patients with 6-month chronic low back pain who were willing to follow patient education manual. Patients were assessed for pain, disability due to backpain and lumbar ranges, at baseline, 2nd, 4th and 6th week of intervention. The SPSS 20.0 version was used to analyse data. Tests of normality were executed that whether data was normative or non-parametric, based on which outcomes were compared either using independent samples t test or Mann-Whitney test.

DETAILED DESCRIPTION:
The goal of current study was to figure out how patient education manual can impact the outcomes, such as decreasing pain and disability and increasing range of lumbar spine, in patients having low back pain. The patient education manual model has been under research in recent time all over the world. There have been mixed results. Mostly there is moderate to high quality evidence in support of patient education that it can help improving the efficacy of physical therapy treatment. However, the previous literature lacks in uniformity of outcome measures used in the studies and spinal ranges have not been studied in majority studies.

This study was conducted by developing a patient education manual given to patients along with routine physical therapy. The study findings showed that the patients with combination of patient education manual and routine physical therapy improved their disability level significantly more than the patients in control group receiving routine physical therapy alone. However, there was no significant difference in improvement of pain itself and spinal ranges of lumbar region except lumbar flexion which was improved significantly among patient education manual group. When the analysis was performed for within group pre and post interventional difference in both groups separately, it was seen that patient improved in both groups significantly at all stages of measurements such as 2nd, 3rd and 6th week, p value less than 0.05.

Looking closer, it was seen that pain was improving similarly in both groups, p value more than 0.05. However, it was slightly better in Group A, having combination of patient education manual and routine physical therapy, with a slight mean difference i.e. -.33333 at 2nd and 4th week and -.41667 at 6th week post intervention. In past studies pain has been reported to be significantly better with patient education groups.

The disability was measured by Oswestry Disability Index for back pain. It was seen that patients having patient education manual significantly improved at all assessment stages i.e. at 2nd, 4th and 6th week, p value less than 0.05. This was the only outcome in this study showing a significantly better effect of patient education manual with straight and clear findings. The mean difference was of 4.25000 at 2nd week, while peak mean difference of 8.83333 points was seen at 4th week which declined to 4.83333 at 6th week but it was still significantly better as compared to routine physical therapy group. It also indicated the gradually fading off difference in long term assessment. In previous studies functional has always been found to improve with patient education. This might due to nature of this outcome which is based on patients' experience and perception, which means due to patient education or information material, it is possible that it has uplifted moral of patients and ultimately, they feel better in all aspects of function. Whatsoever the reason, disability can be greatly improved by use of patient education method in patient with low back pain.

The spinal ranges was the special outcome measure in current study that has been addressed the least in previous literature. It was seen that except lumbar flexion, all ranges were improving without any significant difference, even the improvement in lumbar flexion became same at 6th week assessment. Moreover, there was no consistency in mean difference of ranges, some ranges improved slightly better at one stage of assessment while the same ranges were slightly less improved at other stage, but overall there was no significant difference.

A study had discussed effect of patient education on ranges in terms of its long-term impact and recurrence of hypomobility in spinal region. The study has multiple outcome measures such as pain, disability, ranges and quality of life. The study suggested that all in short term patient education played a significantly better role in improving pain, function and life quality but ranges were no different. Furthermore, all ranges were not measured due to their consistently being similar.

It can be said that all outcomes in which were clinician-based has no difference of improvement in patient education manual group or that of control group while the outcome which were based on patient's perception were improved more among patient education manual group. This pattern can be seen in satisfaction with manual therapy. Although, satisfaction was not associated with treatment group as shown by non-significant p value of chi square more than 0.05, but it can be seen that patients with patient education manual reported themselves to be 'very satisfied' category while in control group the majority patients reported themselves in 'satisfied' category. This showed that all patients were satisfied with care provided for treatment of backpain but providing a patient education manual can further boost their satisfaction which is then reflected in their function.

In short, the outcomes such as function were improved with combination of patient education manual and routine physical therapy while the pain and ranges were no different with or without patient education manual. There needs further studies with more sample size and long term assessment in order see long term impact of patient education manual.

ELIGIBILITY:
Inclusion Criteria:

* 6 months chronic,
* localized low back pain

Exclusion Criteria:

* Patients with radicular low back pain
* Ankylosing spondylitis
* spinal stenosis
* Fibromyalgia
* 0steoprosis
* Cognitive impairment
* Traumatic injury

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 6th Week
  The Oswestry Disability Index (ODI) (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tool. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6th Week
  NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

OTHER OUTCOMES:
GONIOMETER | 6th Week
  A goniometer is a device used in physical therapy to measure the range of motion around a joint in the body. We will use this to measure range of motions ROM on spine, Flexion, Extension, Rotation, Sideflexion R & L

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur-Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Salamat Hospital,Satellite Town, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahin N, Karahan AY, Albayrak I. Effectiveness of physical therapy and exercise on pain and functional status in patients with chronic low back pain: a randomized-controlled trial. Turk J Phys Med Rehabil. 2017 Aug 9;64(1):52-58. doi: 10.5606/tftrd.2018.1238. eCollection 2018 Mar. PMID 31453489
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Background] Traeger AC, Lee H, Hubscher M, Skinner IW, Moseley GL, Nicholas MK, Henschke N, Refshauge KM, Blyth FM, Main CJ, Hush JM, Lo S, McAuley JH. Effect of Intensive Patient Education vs Placebo Patient Education on Outcomes in Patients With Acute Low Back Pain: A Randomized Clinical Trial. JAMA Neurol. 2019 Feb 1;76(2):161-169. doi: 10.1001/jamaneurol.2018.3376. PMID 30398542
- [Background] Pieber K, Herceg M, Quittan M, Csapo R, Muller R, Wiesinger GF. Long-term effects of an outpatient rehabilitation program in patients with chronic recurrent low back pain. Eur Spine J. 2014 Apr;23(4):779-85. doi: 10.1007/s00586-013-3156-z. Epub 2014 Jan 11. PMID 24413743
- [Background] Hanney WJ, Masaracchio M, Liu X, Kolber MJ. The Influence of Physical Therapy Guideline Adherence on Healthcare Utilization and Costs among Patients with Low Back Pain: A Systematic Review of the Literature. PLoS One. 2016 Jun 10;11(6):e0156799. doi: 10.1371/journal.pone.0156799. eCollection 2016. PMID 27285608
- [Background] Medeiros FC, Costa LOP, Added MAN, Salomao EC, Costa LDCM. Longitudinal Monitoring of Patients With Chronic Low Back Pain During Physical Therapy Treatment Using the STarT Back Screening Tool. J Orthop Sports Phys Ther. 2017 May;47(5):314-323. doi: 10.2519/jospt.2017.7199. Epub 2017 Mar 29. PMID 28355979
- [Background] Barbari V, Storari L, Ciuro A, Testa M. Effectiveness of communicative and educative strategies in chronic low back pain patients: A systematic review. Patient Educ Couns. 2020 May;103(5):908-929. doi: 10.1016/j.pec.2019.11.031. Epub 2019 Dec 4. PMID 31839351
- [Background] Beattie PF, Silfies SP, Jordon M. The evolving role of physical therapists in the long-term management of chronic low back pain: longitudinal care using assisted self-management strategies. Braz J Phys Ther. 2016 Nov-Dec;20(6):580-591. doi: 10.1590/bjpt-rbf.2014.0180. Epub 2016 Jun 30. PMID 28001268
- [Background] Burns SA, Cleland JA, Rivett DA, Snodgrass SJ. Effectiveness of physical therapy interventions for low back pain targeting the low back only or low back plus hips: a randomized controlled trial protocol. Braz J Phys Ther. 2018 Sep-Oct;22(5):424-430. doi: 10.1016/j.bjpt.2018.08.014. Epub 2018 Sep 7. PMID 30217693
- [Background] Cherkin DC, Deyo RA, Street JH, Hunt M, Barlow W. Pitfalls of patient education. Limited success of a program for back pain in primary care. Spine (Phila Pa 1976). 1996 Feb 1;21(3):345-55. doi: 10.1097/00007632-199602010-00019. PMID 8742212
- [Background] Davin S, Lapin B, Mijatovic D, Fox R, Benzel E, Stilphen M, Machado A, Katzan IL. Comparative Effectiveness of an Interdisciplinary Pain Program for Chronic Low Back Pain, Compared to Physical Therapy Alone. Spine (Phila Pa 1976). 2019 Dec 15;44(24):1715-1722. doi: 10.1097/BRS.0000000000003161. PMID 31794508
- [Background] de Souza FS, Ladeira CE, Costa LOP. Adherence to Back Pain Clinical Practice Guidelines by Brazilian Physical Therapists: A Cross-sectional Study. Spine (Phila Pa 1976). 2017 Nov 1;42(21):E1251-E1258. doi: 10.1097/BRS.0000000000002190. PMID 28399548
- [Background] Deutscher D, Werneke MW, Hayes D, Mioduski JE, Cook KF, Fritz JM, Woodhouse LJ, Stratford PW. Impact of Risk Adjustment on Provider Ranking for Patients With Low Back Pain Receiving Physical Therapy. J Orthop Sports Phys Ther. 2018 Aug;48(8):637-648. doi: 10.2519/jospt.2018.7981. Epub 2018 May 22. PMID 29787696
- [Background] Du S, Hu L, Dong J, Xu G, Chen X, Jin S, Zhang H, Yin H. Self-management program for chronic low back pain: A systematic review and meta-analysis. Patient Educ Couns. 2017 Jan;100(1):37-49. doi: 10.1016/j.pec.2016.07.029. Epub 2016 Jul 25. PMID 27554077
- [Background] Fritz JM, Kim M, Magel JS, Asche CV. Cost-Effectiveness of Primary Care Management With or Without Early Physical Therapy for Acute Low Back Pain: Economic Evaluation of a Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 Mar;42(5):285-290. doi: 10.1097/BRS.0000000000001729. PMID 27270641